CLINICAL TRIAL: NCT01748942
Title: A Randomized, Placebo Controlled, Double Blinded Study of Corticosteroid Treatment for the Reduction of Postoperative Pain Following Transoral Robotic Surgery
Brief Title: Dexamethasone in Reducing Oral Pain and Dry Mouth After Surgery in Patients With Oropharyngeal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Daniel Clayburgh, Assistant Professor, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00008071; NCI-2012-02780 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CPC-12095-L; CR00021919; IRB00008071 (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Dysphagia; Pain; Stage I Oropharyngeal Squamous Cell Carcinoma; Stage II Oropharyngeal Squamous Cell Carcinoma; Stage III Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Deglutition Disorders; Pain; Squamous Cell Carcinoma of Head and Neck | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (treatment) (Experimental): Patients receive dexamethasone IV at the time of surgery and PO every 8 hours for up to 4 days following surgery.
  Interventions: Drug: Dexamethasone; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Transoral Robotic Surgery
- Arm II (control) (Active Comparator): Patients receive dexamethasone IV at the time of surgery and placebo PO every 8 hours for up to 4 days following surgery.
  Interventions: Drug: Dexamethasone; Other: Placebo; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Transoral Robotic Surgery

INTERVENTIONS:
Drug: Dexamethasone — Given IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
  Arms: Arm I (treatment)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (control)
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Transoral Robotic Surgery — Undergo TORS
  Other Names: TORS

SUMMARY:
This randomized pilot clinical trial studies dexamethasone in reducing oral pain and dry mouth after surgery in patients with oropharyngeal cancer. Dexamethasone may help lower pain and dry mouth caused by surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To prospectively determine if a longer 4-day course of dexamethasone (or equivalent) for the management of postoperative pain and dysphagia following transoral robotic surgery (TORS) is superior to the current standard of a single injection of dexamethasone 10 mg.

SECONDARY OBJECTIVES:

I. Determine the effect of postoperative corticosteroids on postoperative dysphagia following TORS.

II. Determine the effect of postoperative corticosteroids on length of hospital stay following TORS.

III. Determine the complications associated with postoperative corticosteroid use after TORS.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive dexamethasone intravenously (IV) at the time of surgery and orally (PO) every 8 hours for up to 4 days following surgery.

ARM II: Patients receive dexamethasone IV at the time of surgery and placebo PO every 8 hours for up to 4 days following surgery.

After completion of study treatment, patients are followed up for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with oropharyngeal squamous cell carcinoma (SCC) that are surgical candidates
* Macroscopic resection of the tumor via TORS must be planned with curative intent
* Patient must be willing to remain on corticosteroid therapy for 4 days postoperatively
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with known distant metastases or other malignancies
* Patients with a history of allergy or adverse reaction to corticosteroids
* Patients with a history of diabetes
* Patients with fasting capillary blood glucose of > 140 on the day of surgery
* Patients on chronic corticosteroids
* Chronic alcohol abuse (> 6 alcoholic beverages daily)
* Patients with a history of severe chronic pain on high dose narcotics (> 25 mg of oxycodone or equivalent daily) preceding diagnosis of cancer
* Patients taking significant cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors or inducers, i.e. protease inhibitors (ritonavir, nelfinavir, etc), clarithromycin, ketoconazole, fluconazole, verapamil, diltiazem, carbamazepine, phenytoin, phenobarbital, Rifampin, efavirenz, nevirapine
* Patients who have received any investigational medication within 6 weeks of enrollment, or who are scheduled to receive an investigational drug during the course of the study
* Patients who will undergo complex head and neck surgery in addition to the TORS procedure requiring reconstruction with a free flap
* Patients who have had any previous head and neck surgery that has affected swallowing, voice or speech or who have had previous radiation to the head or neck
* Patients who have any confounding medical or neurological conditions that have the potential to affect cognition, speech or swallowing function; i.e. stroke, neurodegenerative disease, neuromuscular movement disorders, head injury, etcetera
* Psychiatric illness/social situations that would limit compliance with study requirements
* Excluded patients will be allowed to participate in the trial on an observational basis only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-12; Primary Completion 2016-07 (Actual); Study Completion 2017-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Clayburgh, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Derived] Clayburgh D, Stott W, Bolognone R, Palmer A, Achim V, Troob S, Li R, Brickman D, Graville D, Andersen P, Gross ND. A randomized controlled trial of corticosteroids for pain after transoral robotic surgery. Laryngoscope. 2017 Nov;127(11):2558-2564. doi: 10.1002/lary.26625. Epub 2017 Aug 29. PMID 28850681

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Treatment) | Arm II (Control)
Started | 39 | 37
Completed | 35 | 33
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Treatment) | Arm II (Control) | Total
Number analyzed (Participants) | 35 | 33 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 28 | 60
  >=65 years | 3 | 5 | 8
Age, Continuous [Mean (Full Range); unit: years] | 56 [44 to 72] | 60 [44 to 75] | 58 [44 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 32 | 29 | 61
Region of Enrollment [Number; unit: participants]
  United States | 35 | 33 | 68
VAS pain score [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Scale (VAS) is a 0-10 scale for patients to indicate intensity level of pain with 0 indicating "No pain" and 10 indicating "Worst possible, unbearable, excruciating pain".
  units on a scale | 1.1 (1.8) | 0.6 (1.3) | 0.9 (1.6)
Tumor stage [Count of Participants; unit: Participants] — Tumor stage is assessed using American Joint Committee on Cancer (AJCC) TNM staging of oropharyngeal squamous cell carcinoma:
  T1 = Tumor 2 cm or less in greatest dimension. T2 = Tumor more than 2 cm but not more than 4 cm in greatest dimension. T3 = Tumor more than 4 cm in greatest dimension or extension to lingual surface of epiglottis.
  T4a = Moderately advanced local disease. T4b = Very advance local disease.
  Participants
    T1 | 21 | 15 | 36
    T2 | 14 | 18 | 32
EAT-10 score [Mean (Standard Deviation); unit: units on a scale] — Mean overall score of the EAT-10 tool. The Eating Assessment Tool (EAT-10) is a 10 item questionnaire that evaluates swallowing and the extent of how problematic with certain eating activities. Questions are answered using a five point (0-4) plus Not Applicable scale with 0 = "No problem" and 4= "Severe problem".
  units on a scale | 5.9 (7.6) | 3.5 (6.2) | 4.6 (6.9)
PSS normalcy of diet [Mean (Standard Deviation); unit: units on a scale] — Performance Status Score (PSS) - Normalcy of Diet score is a 0-100 scale that measures diet restrictions with 0= "Non-oral feeding (tube fed)" and 100 = "Full diet (no restrictions)"
  units on a scale | 92.3 (16.4) | 94.2 (15.0) | 93.8 (15.4)
UM-QOL eating score [Mean (Standard Deviation); unit: units on a scale] — The University of Michigan Head and Neck Quality of Life Questionnaire (UM-QOL) is 20 item, 1-5 scale, questionnaire that measures how much the patient has been bothered during various activities as a result of head and neck condition or treatment in the past four weeks with 1= "Not at all" and 5="Extremely".
  units on a scale | 89.6 (17.8) | 93.75 (12.7) | 89.6 (17.8)

OUTCOME MEASURES:

1. Primary Outcome: Pain Visual Analogue Scale (VAS) Score Measured at 10-point Scale
Description: Visual Analog Scale (VAS) is a 0-10 scale for patients to indicate intensity level of pain with 0 indicating "No pain" and 10 indicating "Worst possible, unbearable, excruciating pain". A descriptive time plot of VAS scores will be produced for all enrolled subjects, with loess curve fitted separately for the experimental and control groups. A linear mixed effects model will be used to compare the pain VAS scores between the experimental and control groups.
Time Frame: 21 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Treatment) | Arm II (Control)
Number analyzed (Participants) | 35 | 33
units on a scale
  Postoperative day #1 | 7.4 (2.0) | 6.8 (2.3)
  Postoperative day #2 | 6.0 (2.0) | 6.4 (2.1)
  Postoperative day #3 | 5.3 (2.0) | 6.7 (1.9)
  Postoperative day #7-21 | 3.0 (1.8) | 2.5 (1.9)
Statistical Analysis 1: Comparison: Arm I (Treatment) vs Arm II (Control); Test type: Superiority; p = 0.25, Mixed Models Analysis

2. Secondary Outcome: Complications Associated With Postoperative Corticosteroid Use After TORS
Description: A descriptive statistical analysis will be conducted on complications.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Treatment) | Arm II (Control)
Number analyzed (Participants) | 35 | 33
Participants
  complication present | 10 | 7
  no complication | 25 | 26

3. Secondary Outcome: Eating Assessment Tool (EAT)-10 Scores
Description: Statistical Analysis between placebo and steroid cohorts to assess differences. The Eating Assessment Tool (EAT-10) is a 10 item questionnaire that evaluates swallowing and the extent of how problematic with certain eating activities. Questions are answered using a five point (0-4) plus Not Applicable scale with 0 = "No problem" and 4= "Severe problem". A descriptive time plot will be produced for EAT-10 scores using baseline and postoperative measurements on days 3 and day 7-21. Descriptive statistical analyses will be conducted for a summary of EAT-10 scores at baseline, days 3 and day 7-21 after surgery. A linear mixed effects model will be used to compare the EAT-10 scores between the two groups.
Time Frame: Up to 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Treatment) | Arm II (Control)
Number analyzed (Participants) | 35 | 33
units on a scale | 20.0 (8.3) | 20.2 (10.7)

4. Secondary Outcome: Length of Hospital Stay (Number of Days Between the Date of Surgery and Date of Discharge)
Description: Kaplan-Meier functions will be fitted to compare the length of hospital stay between the experimental and control groups.
Time Frame: Up to 21 days
Measure: Median (Standard Deviation); unit: days
Arm/Group | Arm I (Treatment) | Arm II (Control)
Number analyzed (Participants) | 35 | 33
days | 5 (1.9) | 4 (1.2)
Statistical Analysis 1: Comparison: Arm I (Treatment) vs Arm II (Control); Test type: Superiority; p < 0.001, Log Rank

5. Secondary Outcome: PSS Normalcy of Diet
Description: Performance Status Score (PSS) - Normalcy of Diet score is a 0-100 scale that measures diet restrictions with 0= "Non-oral feeding (tube fed)" and 100 = "Full diet (no restrictions)"
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Treatment) | Arm II (Control)
Number analyzed (Participants) | 35 | 33
units on a scale | 51.7 (24.4) | 36.7 (23.4)
Statistical Analysis 1: Comparison: Arm I (Treatment) vs Arm II (Control); Test type: Superiority; p = 0.009, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Opioid Use
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: mg of oxycodone equivalent
Arm/Group | Arm I (Treatment) | Arm II (Control)
Number analyzed (Participants) | 35 | 33
mg of oxycodone equivalent | 137.1 (115.2) | 147.3 (90.4)
Statistical Analysis 1: Comparison: Arm I (Treatment) vs Arm II (Control); Test type: Superiority; p = 0.33, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: UM-QOL Eating
Description: The University of Michigan Head and Neck Quality of Life Questionnaire (UM-QOL) is 20 item, 1-5 scale, questionnaire that measures how much the patient has been bothered during various activities as a result of head and neck condition or treatment in the past four weeks with 1= "Not at all" and 5="Extremely". The scores are calculated using a Likert Scale, which transforms the 1-5 choices into a 0-100 scale with 100 being normal and 0 being poor quality of life. This test contains separate domains (eating, etc.) that can be scored independently. Scores were analyzed between cohorts pre and post operatively.
Time Frame: 21 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Treatment) | Arm II (Control)
Number analyzed (Participants) | 35 | 33
units on a scale | 59.3 (19.5) | 60.1 (19.4)
Statistical Analysis 1: Comparison: Arm I (Treatment) vs Arm II (Control); Test type: Superiority; p = 0.96, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Days With Feeding Tube
Time Frame: 12 months
Measure: Median (Full Range); unit: days
Arm/Group | Arm I (Treatment) | Arm II (Control)
Number analyzed (Participants) | 35 | 33
days | 4 [2 to 311] | 11 [2 to 298]
Statistical Analysis 1: Comparison: Arm I (Treatment) vs Arm II (Control); Test type: Superiority; p = 0.15, Log Rank

ADVERSE EVENTS:
Arm/Group | Arm I (Treatment) | Arm II (Control)
Serious Adverse Events (participants affected / at risk) | 10/35 | 7/33
Other Adverse Events (participants affected / at risk) | 0/35 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Treatment) (N=35) | Arm II (Control) (N=33)
oropharyngeal hemorrhage (Surgical and medical procedures) | 4 | 3 (3)
Neck hematoma (Surgical and medical procedures) | 2 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Chyle leak (Surgical and medical procedures) | 1 | 0
Readmission/failure to thrive (Surgical and medical procedures) | 2 | 0
abscess (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes